CLINICAL TRIAL: NCT05353530
Title: Phase I Study -To Assess Safety and Feasibility of IL-8 Receptor Modified Patient-derived Activated CD70 CAR T Cell Therapy in CD70+ Adult GBM and Pediatric High-Grade Gliomas (pHGG)
Brief Title: IL-8 Receptor-modified CD70 CAR T Cell Therapy in CD70+ Adult Glioblastoma
Acronym: IMPACT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: AM Rosen Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202200057-A; OCR41673 (Other: University of Florida)
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma Multiforme; Glioblastoma
Keywords: CAR T Cell; Brain Tumor; Brain Cancer; Glioblastoma Multiforme; Immunotherapy
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Receptors, Interleukin-8B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 8R-70CAR T cells (Experimental): Cohort 1 will receive 1 x 10^6 cells/kg. Cohort 2 will receive 1 x 10^7 cells/kg. Cohort 3 will receive 1 x 10^8 cells/kg. Cohort 4 will receive Cy/Flu + CAR T cells at established maximum tolerated dose.
  Interventions: Biological: Ex-Vivo expanded autologous IL-8 receptor (CXCR2) modified CD70 CAR (8R-70CAR) T cells

INTERVENTIONS:
Biological: Ex-Vivo expanded autologous IL-8 receptor (CXCR2) modified CD70 CAR (8R-70CAR) T cells — Single dose of 8R-70CAR T cells administered IV
  Other Names: 8R-70CAR T cells

SUMMARY:
This is a phase I study to assess the safety and feasibility of IL-8 receptor modified patient-derived activated CD70 CAR T cell therapy in CD70+ adult glioblastoma

DETAILED DESCRIPTION:
Newly diagnosed CD70 positive adult GBM patients who have undergone surgery for maximal debulking will be enrolled in this 3+3 design dose-escalation clinical trial and undergo peripheral venipuncture for collection of PBMCs for generation of investigational 8R-70CAR T Cell vaccine. Patients will then undergo standard of care chemoradiation. Immunotherapy will begin 2 weeks (-7/+4 days) after completion of radiation. One single dose of 8R-70CAR T cells will be administered IV. The dose will depend on the enrolling cohort. Dose escalation will follow the traditional 3+3 design.

ELIGIBILITY:
Inclusion Criteria (Adult GBM):

* Age ≥ 18 years
* Newly-diagnosed de novo GBM based on the absence of previous history of brain tumor (WHO Grade IV glioma) by histopathology or molecular studies. (secondary GBM not eligible)
* The tumor must have a supratentorial component
* CD70 positive (≥5%, 1+)

Tumor expression will be scored on a scale of 0 to 3 staining intensity:

0 = Negative

1. = Low level
2. = Moderate level
3. = High level

   * The criteria for inclusion will be at least 5% of the cells scoring 1+ staining intensity (> 5%, 1+).

     * Surgical resection of tumors with less than 3cm x 3cm (9 cm2) residual enhancing tumor as a product of longest perpendicular planes by MRI or biopsy only for tumor measuring less than 3cm x 3cm
     * Karnofsky Performance Status (KPS) of > 70%
     * CBC with differential with adequate bone marrow function as defined below:
   * Absolute neutrophil count (ANC) ≥ 1500 cells/mm3.
   * Platelet count ≥ 100,000 cells/mm3.
   * Hemoglobin ≥ 10 g/dl. (The use of transfusion or other intervention to achieve Hgb ≥ 10 g/dl is acceptable.)

     • Adequate renal function as defined below:
   * BUN ≤ 25 mg/dl
   * Creatinine ≤ 1.7 mg/dl

     • Adequate hepatic function as defined below:
   * Bilirubin ≤ 2.0 mg/dl
   * ALT ≤ 5 times institutional upper limits of normal for age
   * AST ≤ 5 times institutional upper limits of normal for age

     * Signed informed consent. If the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the legally authorized representative.
     * For females of childbearing potential, a negative serum pregnancy test at enrollment.
     * Women of childbearing potential (WOCBP) must be willing to use an acceptable contraceptive method to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug.
     * Males with female partners of childbearing potential must agree to practice adequate contraceptive methods throughout the study and should avoid conceiving children for 24 weeks following the last dose of study drug.

Exclusion Criteria (Adult GBM):

* Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3years. (In situ cancer are permissible)
* Metastases detected below the tentorium or beyond the cranial vault
* Leptomeningeal disease beyond the cranial vault. (Focal, adjacent and leptomeningeal involvement is allowable at the discretion of the PI).
* Recurrent or multifocal malignant gliomas.
* The patient is not a candidate for cellular therapy as assessed by the study bone marrow transplant physician.
* Known immunosuppressive disease or human immunodeficiency virus (HIV) infection.

Rationale: The need to exclude patients with the immunosuppressive disease or human

* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization.
  * Transmural myocardial infarction within the last 6 months.
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the initiation of XRT/TMZ.
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the initiation of XRT/TMZ.
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
  * Patients with an autoimmune disease requiring medical management with immunosuppressants.
  * Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy.
  * Active connective tissue disorders such as lupus or scleroderma that, in the investigator's opinion, place the patient at high risk for radiation toxicity.
* Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant.
* Patients treated on any other therapeutic clinical protocols within 30 days prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2042-12 (Estimated)

PRIMARY OUTCOMES:
Safety of 8R-70CAR T-cell therapy in adult patients with de novo CD70+ GBM | 28 days post-infusion
  Defined as ≤ 1 DLT out of 6 patients is observed at the 1x10^8 cells/Kg dose. Dose-Limiting toxicity (DLT) will be defined as any adverse event attributable (possible, probable, or definite) to the administration of 8R-70CAR T cells and occurring from the time of infusion through 28 days post-infusion.
Feasibility of 8R-70CAR T-cell therapy in adult patients with de novo CD70+ GBM | 10 weeks
  Feasibility will be defined as the ability to infuse 8R-70CAR T-cell safely in 66.7 % of enrolled patients (patients who signed consent and were deemed eligible for the study).

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Ghiaseddin, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No